CLINICAL TRIAL: NCT03061786
Title: Prognosis of Acute Kidney Injury:China Collaborative Study on AKI（CCS-AKI）Study
Status: Recruiting | Type: Observational
Sponsor: XinLing Liang (Other)
Responsible Party: Sponsor-Investigator, XinLing Liang, Director of Division of Nephrology and Blood Purification Center of Guangdong General Hospital, Guangdong Provincial People's Hospital
Organization: Guangdong Provincial People's Hospital (Other)
Other Study IDs: CCS-AKI P2011-2016
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- AKI
- non-AKI

SUMMARY:
Acute kidney injury (AKI) is a common clinical syndrome, especially in the hospital patients. AKI is recognized as an important risk factor for incident chronic kidney disease, accelerated progression to end-stage renal disease,and increased risk of short-term and long-term mortality.This study is to observe the prognosis of hospitalized patients with AKI in China.

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed with acute kidney injury, according to KDIGO criteria

Exclusion Criteria:

* Nephrectomy
* Kidney transplantation
* Peak serum creatinine of less than 53µ mol/L
* Serum creatinine decrease after amputation
* Patients died during hospitalization
* End-stage kidney disease(chronic kidney disease stage 5)
* malnutrition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients
Sampling Method: Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2017-01; Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
estimated glomerular filtration rate decline | 2 years
  >50% baseline
Chronic kidney disease classification upgrade | 5 years
New cardiovascular events | 5 years
All-cause mortality | 5 years

SECONDARY OUTCOMES:
AKI recovery | 5 years
Rehospitalization | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China